CLINICAL TRIAL: NCT02071836
Title: A Web Application to Reduce Heavy Drinking in First-time DWI Offenders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Behavior Therapy Associates, LLP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NIAAA 2R44020174
Record Dates: First submitted 2014-02-24; First posted 2014-02-26 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2016-09

CONDITIONS: Driving While Intoxicated; Driving Under the Influence; Heavy Drinking; Alcohol Abstinence
Keywords: web application; DWI intervention; DUI intervention; Experimental group: Right Turns + treatment as usual; Control group: Treatment as usual
MeSH Terms: conditions — Driving Under the Influence; Alcohol Abstinence | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Right Turns web application (Experimental): Right Turns web application
  Interventions: Behavioral: Right Turns web application; Behavioral: Treatment as usual
- Treatment as usual (Active Comparator): Treatment as usual
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Right Turns web application
  Arms: Right Turns web application
Behavioral: Treatment as usual

SUMMARY:
The overall objective of this project is to develop, evaluate, and disseminate a web application for first-time DWI offenders that will provide them with an age-appropriate brief motivational intervention (BMI) to motivate them to reduce their drinking and a cognitive behavioral intervention (CBI) for to help them achieve and maintain abstinence. The goal is to reduce heavy drinking and consequently the risk for future drunk driving.

The specific objectives of this Phase II are:

* Completing the development of the Right Turns prototype based on feedback from the Phase I pilot study participants. This includes: providing more structure and guidance as participants work in the Tool Box section of the program; simplifying the content of the Tool Box; further R&D in the text messaging feature for 2nd and 3rd tier cellular providers; implement a customized pdf report function for progress reports from the program to users' probation officers (under control of the user); developing a follow-up component and outcome reports; and revising the videos in the Tool Box to reflect greater diversity and a younger population of drinkers.
* Conducting a randomized clinical trial of the program with first time DWI/DUI offenders who are recruited locally, collecting follow-up data, analyzing the data, and reporting the results.

ELIGIBILITY:
Inclusion Criteria:

* be a first-time DWI offender
* have a 5th grade reading level
* has a computer with Internet access at home
* own a cell phone with text messaging

Exclusion Criteria:

* age less than 18
* recent history of uncontrolled psychotic or bipolar behavior
* evidence of significant cognitive impairment from brain dysfunction (e.g., head injury)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Quantity/frequency of alcohol use: Form 90 | 3 months
  Quantity/frequency of drinking in previous 3 months
Inventory of Drug Use Consequences (InDuC) | 3 months
  Quantity/frequency of alcohol and drug related problems in the previous 3 months

SECONDARY OUTCOMES:
Self-efficacy | at enrollment
  The Alcohol Abstinence Self-Efficacy scale measures one's confidence in remaining abstinent in various situations.

CONTACTS AND LOCATIONS:
Overall Officials: Reid K Hester, Ph.D., Principal Investigator — Behavior Therapy Associates, LLC
Locations (1):
- Behavior Therapy Associates, LLC, Albuquerque, New Mexico, United States